CLINICAL TRIAL: NCT03552926
Title: Constitution of a Clinico-radiological Database and a Biobank for Patients With Lacunar Infarcts at Lariboisière Fernand-Widal and Sainte Anne Hospitals
Brief Title: Constitution of a Clinico-radiological Database and a Biobank for Patients With Lacunar Infarcts
Acronym: DHU-LAC
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P150602
Record Dates: First submitted 2018-03-27; First posted 2018-06-12 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Lacunar Strokes
Keywords: Small subcortical infarct; Cerebrovascular disorders; Neurocognitive and cardiovascular disorders; Disability; Dementia; Stroke
MeSH Terms: conditions — Stroke, Lacunar; Cerebrovascular Disorders; Cardiovascular Diseases; Dementia; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine in patients with a recent lacunar strokes (<15 days), the natural history of cognitive disturbances and disability.

DETAILED DESCRIPTION:
This bi-centric cohort study aims at determining in patients with recent lacunar strokes (<15 days), the main clinical, radiological, or genetic predictive markers of recurrent stroke, cognitive impairment, dementia, depression gait disturbances and disability.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* History of recent (less than 15 days) neurological deficit related to a small subcortical infarct (evidenced by medical history or physical examination)
* Diagnosis of recent small subcortical infarct on MRI (hyperintensity on diffusion-weighted imaging showing an infarction in the territory of one perforating artery) presumably responsible for the corresponding neurological deficit
* Lesion diameter mess than 20 mm
* Ability to comply with scheduled follow-up and annual neurological evaluation
* Affiliation to the national French health insurance (sécurité sociale)
* Signature of informed consent

Exclusion Criteria:

* Prior diagnosis of dementia according to DSM IV criteria
* Prior severe disability with Rankin scale ≥ 4
* Serious concomitant systemic disorder that can compromise the follow-up study;
* Leukoencephalopathy of non-vascular origin;
* Severe psychiatric disorder;
* Inability to obtain an informed signed consent from the patient or his/her family;
* Medical contraindication or refusal to undergo cerebral magnetic resonance scanning (MRI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recent small subcortical infarct (less than 15 days) evaluated as outpatient or inpatient in the Neurology Departments at the Hospital Lariboisière Fernand-Widal or at the Centre Hospitalier Sainte-Anne in Paris
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-06-06 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Time to the occurrence of cognitive decline | 5 years
  diagnosis of mild or major neurocognitive disorder according to DSM5

SECONDARY OUTCOMES:
Recurrent stroke | 5 years
  Time to the occurrence of one of the following event
Dementia | 5 years
  diagnosis of major neurocognitive disorder (dementia) according to DSMV criteria
Transient ischaemic attacks | 5 years
  " Transient ischemic attack " is a well recognized outcome in clinical trials in neurovascular disorders. We chose the most commonly definition of TIA according to international guidelinesorigin, without recent ischemic lesion on diffusion weighted imaging
Cardiovascular events | 5 years
  myocardial infarction or cardiac failure
Attacks of migraine with aura | 5 years
  according to international classification of headache disorders 2nd edition (ICHD-2)
Memory complaints | 5 years
  any spontaneous complain of memory deficit, irrespective of the neuropsychological battery results
Depression or other mood alterations | 5 years
  " HADS refers to Hamilton Anxiety and Depression Scale, as stated initially in the title. The scale comprises 14 questions with structured answers ranging from 0 to 3, leading to 2 scores (1 for anxiety, 1 for depression, ranging each from 0 to 21). In each case, larger values are considered to represent worse outcomes. Scores larger or equal to 11 correspond to thresholds to define anxiety and depression "
Behavioural disorders | 5 years
  according to DSMV classification
Balance disturbances | 5 years
  according to the SPPB battery
Falls | 5 years
  according to patient's relatives recording
Urinary complaints | 5 years
  any spontaneous complain from the patients and/or his relative

CONTACTS AND LOCATIONS:
Overall Officials: Eric JOUVENT, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Lariboisière, Paris, France

REFERENCES:
- [Derived] Grosset L, Dimitrovic A, Guillonnet A, Tamazyan R, Benzakoun J, Dusonchet A, Chabriat H, Oppenheim C, Zuber M, Calvet D, Jouvent E. MRI-Proven Incident Ischemia: A New Marker of Disease Progression in Small Vessel Diseases. Stroke. 2025 Jan;56(1):39-45. doi: 10.1161/STROKEAHA.124.048046. Epub 2024 Nov 21. PMID 39569496